CLINICAL TRIAL: NCT04381949
Title: Interest of Tracheal Extubation in Positive Pressure on Postoperative Oxygenation in Adult Digestive Surgery: Prospective Randomized Study
Brief Title: Interest of Tracheal Extubation in Positive Pressure on Postoperative Oxygenation in Adult Digestive Surgery: Prospective Randomized Study ExPress
Acronym: ExPress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019/0351/HP
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Patients Undergoing Digestive Surgery With Orotracheal Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard extubation Arm (No Intervention)
- Positive pressure extubation arm (Experimental)
  Interventions: Procedure: positive pressure extubation

INTERVENTIONS:
Procedure: positive pressure extubation — Two arms:
  the first with "classic" extubation with disconnection of the ventilator and the second with an extubation without disconnection of the respiratory "positive pressure"
  Arms: Positive pressure extubation arm

SUMMARY:
Evaluation of a postoperative tracheal extubation protocol under positive pressure in accordance with international recommendations.

Two arms: the first with "classic" extubation with disconnection of the respirator and the second with extubation without disconnection of the respiratory, as recommended.

Computer Randomization with a 1: 1 ration

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 and <80
* Patient going to benefit from general anesthesia with orotracheal intubation for surgery lasting more than 60 minutes at the visceral surgery unit of the Rouen University Hospital.
* Person affiliated to a social security scheme
* Person who has read and understood the newsletter and signed the consent form

Exclusion Criteria:

* Minor patients or age> 80 years
* History of Obstructive Sleep Apnea Syndrome
* Chronic respiratory failure / History of chronic obstructive pulmonary disease
* Surgery < 60 minutes
* Use of methylene blue intraoperatively
* Extubation finally performed in the operating room
* orotracheal intubation difficult to induce general anesthesia
* Suspected inhalation during orotracheal intubation
* Pneumothorax per operative
* Heart failure authenticated by trans thoracic ultrasound <50%
* Neuromuscular pathologies (myasthenia gravis, myopathies)
* Body mass index> 35
* Emergency surgery
* Patient with an ASA IV score (ie according to the definition of the American Society of Anesthesiology)
* Major surgical complications (hemorrhagic shock)
* Major anesthetic complications (anaphylactic shock, bronchospasm)
* Pregnant or parturient or lactating woman or woman of childbearing age without proven contraception
* Person deprived of their liberty by an administrative or judicial decision or person placed under the protection of justice / guardianship or curatorship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Desaturation rate | within one hour of tracheal extubation
  defined by a SpO2 < 92%